CLINICAL TRIAL: NCT00103857
Title: A Multicenter, Randomized, Double-Blind Factorial Study of the Co-Administration of MK0431 and Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: MK0431 (Sitagliptin) and Metformin Co-Administration Factorial Study in Patients With Type 2 Diabetes Mellitus (0431-036)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-036; MK0431-036; 2005_003
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Results first posted 2009-05-19 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental): MK0431 100 mg q.d.
  Interventions: Drug: Comparator: MK0431 100 mg q.d. (q.d. = once daily)
- 2 (Active Comparator): Metformin 500 mg b.i.d.
  Interventions: Drug: Comparator: Metformin 500 mg b.i.d.
- 3 (Active Comparator): Metformin 1000 mg b.i.d.
  Interventions: Drug: Comparator: Metformin 1000 mg b.i.d.
- 4 (Experimental): Coadministration of MK0431 and Metformin 50/500 mg b.i.d.
  Interventions: Drug: Comparator: MK0431 50 mg b.i.d. (b.i.d. = twice daily); Drug: Comparator: Metformin 500 mg b.i.d.
- 5 (Experimental): Coadministration of MK0431 and Metformin 50/1000 mg b.i.d.
  Interventions: Drug: Comparator: MK0431 50 mg b.i.d. (b.i.d. = twice daily); Drug: Comparator: Metformin 1000 mg b.i.d.
- 6 (Placebo Comparator): Placebo/Metformin 1000 mg b.i.d.
  Interventions: Drug: Comparator: Placebo (Phase A)/Metformin (Phase B)
- 7 (Experimental): Non-Randomized, Open-Label: Coadministration MK0431 and Metformin 50/1000 mg b.i.d.
  Interventions: Drug: Comparator: Open-Label MK0431/Metformin 50/1000 mg b.i.d.

INTERVENTIONS:
Drug: Comparator: MK0431 50 mg b.i.d. (b.i.d. = twice daily) — MK0431 oral tablets will be started on Day 1 at 50 mg q.d. (q.d. = once daily) and increased after one week to a stable dose of 50 mg b.i.d. (b.i.d. = twice daily) Patients will continue to take MK0431 50 mg b.i.d. for the remainder of the 54-week base study (including the 24-week placebo-controlled Phase A and 30-week active-controlled Phase B) and during the 50-week extension study (for patients who complete the 54-week base study and enter the 50-week extension study) for a total treatment duration of up to 104 weeks.
  Other Names: MK0431
  Arms: 4; 5
Drug: Comparator: MK0431 100 mg q.d. (q.d. = once daily) — MK0431 oral tablets will be started on Day 1 as two 50 mg tablets (100 mg q.d.) (q.d. = once daily) and continued at this dose throughout the 54-week base study (including the 24-week placebo-controlled Phase A and 30-week active-controlled Phase B) and the 50-week extension study (for patients who complete the 54-week base study and enter the 50-week extension study) for a total treatment duration of up to 104 weeks.
  Arms: 1
Drug: Comparator: Placebo (Phase A)/Metformin (Phase B) — During the placebo-controlled period (Day 1 through Week 24/Phase A), metformin and MK0431 matching placebos will be dispensed as oral tablets. At the beginning of the 30-week active-controlled period (Phase B), metformin will be started as 500 mg q.d. (q.d. = once daily) and up-titrated in 500 mg weekly increments to a stable dose of 1000 mg b.i.d. Patients who complete the 54-week base study and who enter the 50-week extension study will continue to take metformin 1000 mg b.i.d. (b.i.d. = twice daily) for a total placebo/metformin treatment duration of up to 104 weeks.
  Arms: 6
Drug: Comparator: Metformin 500 mg b.i.d. — Metformin oral tablets will be started on Day 1 at 500 mg q.d. (q.d. = once daily) and increased after 1 week to a stable dose of 500 mg b.i.d. (b.i.d. = twice daily) Patients will continue to take metformin 500 mg b.i.d. for the remainder of the 54-week base study (including the 24-week placebo-controlled Phase A and 30-week active-controlled Phase B) and during the 50-week extension study (for patients who complete the 54-week base study and enter the 50-week extension study) for a total treatment duration of up to 104 weeks.
  Arms: 2; 4
Drug: Comparator: Open-Label MK0431/Metformin 50/1000 mg b.i.d. — MK0431 oral tablets will be started on Day 1 at 50 mg q.d. (q.d. = once daily) and increased after one week to a stable dose of 50 mg b.i.d. (b.i.d. = twice daily) Metformin oral tablets will be started on Day 1 at 500 mg q.d. and increased by increments of 500 mg per week to achieve a stable dose of 1000 mg b.i.d. The open-label treatment period is 24 weeks.
  Arms: 7
Drug: Comparator: Metformin 1000 mg b.i.d. — Metformin oral tablets will be started on Day 1 at 500 mg q.d. (q.d. = once daily) and increased by increments of 500 mg per week to achieve a stable dose of 1000 mg b.i.d. (b.i.d. = twice daily) Patients will continue to take metformin 1000 mg b.i.d. for the remainder of the 54-week base study (including the 24-week placebo-controlled Phase A and 30-week active-controlled Phase B) and during the 50-week extension study (for patients who complete the 54-week base study and enter the 50-week extension study) for a total treatment duration of up to 104 weeks.
  Arms: 3; 5

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an investigational drug in patients with Type 2 Diabetes Mellitus (T2DM) (a specific type of diabetes).

ELIGIBILITY:
Inclusion Criteria:

54-Week Base Study:

* Patients between the ages of 18 and 78 with Type 2 Diabetes Mellitus (a specific type of diabetes)

  50-Week Extension Study:
* Patients who complete the 54-week base study are eligible to enter the 50-week extension study

Exclusion Criteria:

* Patients who do not have Type 2 Diabetes Mellitus (a specific type of diabetes)

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2005-03-17 (Actual); Primary Completion 2006-07-25 (Actual); Study Completion 2008-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Goldstein BJ, Feinglos MN, Lunceford JK, Johnson J, Williams-Herman DE; Sitagliptin 036 Study Group. Effect of initial combination therapy with sitagliptin, a dipeptidyl peptidase-4 inhibitor, and metformin on glycemic control in patients with type 2 diabetes. Diabetes Care. 2007 Aug;30(8):1979-87. doi: 10.2337/dc07-0627. Epub 2007 May 7. PMID 17485570
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 01-Apr-2005
  Last Patient Last Visit: 29-Feb-2008
  140 study centers worldwide
Pre-assignment Details: Patients 18-78 years with T2DM and an HbA1c 7.5-11% on diet/exercise were eligible for randomization into the 54-week (wk) base study. Patients with an HbA1c >11% or glucose >280 mg/dL were eligible to participate in the Open-label Cohort through Wk 24. Randomized patients who completed the base study were eligible to enter a 50-wk extension study.
Groups:
- Sitagliptin 100 mg q.d.: The Sitagliptin 100 mg q.d. (q.d. = once daily) group includes data from patients randomized to receive treatment with two 50 mg oral tablets of sitagliptin once daily for up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study). Note: In this double-blind, double-dummy study, randomized patients in the base study received a total of 7 tablets (active or placebo) per day administered in the specified tablet images as follows: sitagliptin 50 mg 2 tablets in the morning and 1 tablet in the evening, metformin 500 mg 2 tablets b.i.d. (b.i.d. = twice daily). In the extension study, patients received a total of 7 tablets (active or placebo) per day. Tablets in the image of sitagliptin (active or placebo) were administered as sitagliptin 100 mg 1 tablet in the morning and sitagliptin 50 mg 1 tablet b.i.d. Metformin administration occurred in the same manner as specified in the base study.
- Metformin 500 mg b.i.d.: The Metformin 500 mg b.i.d. (b.i.d. = twice daily) group includes data from patients randomized to receive treatment with oral tablets of metformin 500 mg b.i.d. Treatment was administered as 500 mg q.d. (q.d. = once daily) beginning at randomization/Day 1 and increased after 1 week to a stable dose of 500 mg b.i.d. Patients in this group continued to take metformin 500 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Metformin 1000 mg b.i.d.: The Metformin 1000 mg b.i.d. (b.i.d. = twice daily) group includes data from patients randomized to receive treatment with oral tablets of metformin 1000 mg b.i.d. Treatment was administered as 500 mg q.d. (q.d. = once daily) beginning at randomization/Day 1 and increased over 4 weeks by increments of 500 mg per week to a stable dose of 1000 mg b.i.d. Patients in this group continued to take metformin 1000 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d.: The Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. (b.i.d. = twice daily) group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 50 mg b.i.d + metformin 500 mg b.i.d. Treatment was co-administered as sitagliptin 50 mg q.d. (q.d. = once daily) and metformin 500 mg q.d. beginning at randomization/Day 1; after 1-week, the dose of sitagliptin was increased to 50 mg b.i.d. and the dose of metformin was increased to 500 mg b.i.d. Patients in this group continued to take sitagliptin 50 mg b.i.d. and metformin 500 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d.: The Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. (b.i.d. = twice daily) group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 50 mg b.i.d + metformin 1000 mg b.i.d. Treatment was co-administered as sitagliptin 50 mg q.d. (q.d. = once daily) and metformin 500 mg q.d. beginning at randomization/Day 1; the dose of sitagliptin was increased after 1-week to 50 mg b.i.d and the dose of metformin was increased over 4 weeks by increments of 500 mg per week to 1000 mg b.i.d. Patients in this group continued to take sitagliptin 50 mg b.i.d. and metformin 1000 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Placebo/Metformin 1000 mg b.i.d.: The Placebo/Metformin 1000 mg b.i.d. group (b.i.d. = twice daily) includes data from patients randomized to receive the sequence of treatment with oral tablets of placebo (randomization/Day 1 through Week 24) followed by metformin. Beginning at Week 24, patients were switched in a blinded manner to active treatment with metformin administered as 500 mg q.d. (q.d. = once daily) increased over 4 weeks by increments of 500 mg per week to a stable dose of 1000 mg b.i.d. Patients in this group continued to take metformin 1000 mg b.i.d for the remainder of the up to 30-week Phase B base study treatment period and during the extension study of up to 50 weeks.
- Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC: The Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. (b.i.d. = twice daily) OLC (Open-label Cohort) includes data from non-randomized patients assigned to receive treatment with open-label, oral tablets of sitagliptin and metformin. Treatment was co-administered as sitagliptin 50 mg q.d. (q.d. = once daily) and metformin 500 mg q.d. beginning on Day 1. The dose of sitagliptin was increased after 1-week to 50 mg b.i.d and the dose of metformin was increased over 4 weeks by increments of 500 mg per week to 1000 mg b.i.d. Patients continued to take open-label sitagliptin 50 mg b.i.d. and metformin 1000 mg b.i.d for the remainder of the Phase A treatment period of up to 24 weeks. Results presented for the OLC are through Week 24. Patients in the OLC completed the study at Week 24.
Period: 54-Week Base Study
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC
Started | 179 | 182 | 182 | 190 | 182 | 176 | 117 (Results for the OLC are through Week 24. Results for the 6 randomized groups are through Week 54.)
Completed | 122 | 126 | 135 | 148 | 141 | 115 | 79
Not Completed | 57 | 56 | 47 | 42 | 41 | 61 | 38
Not completed — Adverse Event | 12 | 9 | 11 | 6 | 5 | 11 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 11 | 14 | 8 | 4 | 3 | 14 | 19
Not completed — Lost to Follow-up | 5 | 4 | 7 | 5 | 10 | 9 | 3
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 6 | 4 | 2 | 4 | 0 | 3 | 3
Not completed — Withdrawal by Subject | 17 | 16 | 16 | 15 | 10 | 15 | 4
Not completed — protocol discontinuation criteria | 2 | 5 | 2 | 6 | 5 | 3 | 5
Not completed — patient moved | 0 | 1 | 1 | 2 | 3 | 1 | 0
Not completed — non-compliance with study procedures | 1 | 2 | 0 | 0 | 0 | 2 | 0
Not completed — patient incarcerated | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — laboratory reporting error | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — site error | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — patient intolerance to rescue therapy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: 50-Week Extension Study
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC
Started | 103 (19 randomized patients completed Period 1 but did not enter Period 2.) | 107 (19 randomized patients completed Period 1 but did not enter Period 2.) | 121 (14 randomized patients completed Period 1 but did not enter Period 2.) | 134 (14 randomized patients completed Period 1 but did not enter Period 2.) | 122 (19 randomized patients completed Period 1 but did not enter Period 2.) | 98 (17 randomized patients completed Period 1 but did not enter Period 2.) | 0
Completed | 65 | 80 | 95 | 98 | 101 | 78 | 0
Not Completed | 38 | 27 | 26 | 36 | 21 | 20 | 0
Not completed — Adverse Event | 2 | 3 | 2 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 26 | 15 | 13 | 16 | 8 | 8 | 0
Not completed — Lost to Follow-up | 4 | 0 | 1 | 4 | 3 | 3 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 2 | 8 | 3 | 3 | 0
Not completed — protocol discontinuation criteria | 2 | 2 | 3 | 2 | 3 | 3 | 0
Not completed — non-compliance with study procedures | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — patient moved | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — patient scheduled for elective surgery | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — reason unspecified | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC | Total
Number analyzed (Participants) | 179 | 182 | 182 | 190 | 182 | 176 | 117 | 1208
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.2) | 53.4 (10.2) | 53.2 (9.6) | 54.1 (10.0) | 53.3 (9.6) | 53.6 (10.0) | 52.6 (10.0) | 53.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 93 | 100 | 85 | 105 | 83 | 50 | 602
  Male | 93 | 89 | 82 | 105 | 77 | 93 | 67 | 606
Race/Ethnicity, Customized [Number; unit: participants]
  White | 93 | 87 | 106 | 102 | 95 | 81 | 44 | 608
  Black | 11 | 12 | 9 | 13 | 14 | 17 | 9 | 85
  Hispanic | 52 | 55 | 39 | 55 | 49 | 47 | 54 | 351
  Asian | 6 | 14 | 10 | 9 | 11 | 12 | 1 | 63
  Other | 17 | 14 | 18 | 11 | 13 | 19 | 9 | 101
HbA1c (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 8.9 (1.0) | 8.9 (1.0) | 8.7 (0.9) | 8.8 (1.0) | 8.7 (0.9) | 8.7 (1.0) | 11.2 (1.2) | 9.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 24
Description: HbA1c is measured as a percent. This change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last observed measurement was carried forward to Week 24. The Open-label Cohort group was excluded from the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Metformin 500 mg b.i.d.: The Metformin 500 mg b.i.d. (b.i.d. = twice daily.) group includes data from patients randomized to receive treatment with oral tablets of metformin 500 mg b.i.d. Treatment was administered as 500 mg q.d. (q.d. = once daily) beginning at randomization/Day 1 and increased after 1 week to a stable dose of 500 mg b.i.d. Patients in this group continued to take metformin 500 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Metformin 1000 mg b.i.d.: The Metformin 1000 mg b.i.d. (b.i.d. = twice daily.) group includes data from patients randomized to receive treatment with oral tablets of metformin 1000 mg b.i.d. Treatment was administered as 500 mg q.d. (q.d. = once daily) beginning at randomization/Day 1 and increased over 4 weeks by increments of 500 mg per week to a stable dose of 1000 mg b.i.d. Patients in this group continued to take metformin 1000 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d.: The Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. (b.i.d. = twice daily.) group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 50 mg b.i.d + metformin 500 mg b.i.d. Treatment was co-administered as sitagliptin 50 mg q.d. (q.d. = once daily)and metformin 500 mg q.d. beginning at randomization/Day 1; after 1-week, the dose of sitagliptin was increased to 50 mg b.i.d. and the dose of metformin was increased to 500 mg b.i.d. Patients in this group continued to take sitagliptin 50 mg b.i.d. and metformin 500 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d.: The Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. (b.i.d. = twice daily.) group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 50 mg b.i.d + metformin 1000 mg b.i.d. Treatment was co-administered as sitagliptin 50 mg q.d. (q.d. = once daily) and metformin 500 mg q.d. beginning at randomization/Day 1; the dose of sitagliptin was increased after 1-week to 50 mg b.i.d and the dose of metformin was increased over 4 weeks by increments of 500 mg per week to 1000 mg b.i.d. Patients in this group continued to take sitagliptin 50 mg b.i.d. and metformin 1000 mg b.i.d for the remainder of the treatment period of up to 104 weeks (including the 54-week base study [24-week, placebo-controlled Phase A and 30-week, active-controlled Phase B] and 50-week extension study).
- Placebo/Metformin 1000 mg b.i.d.: The Placebo/Metformin 1000 mg b.i.d. group (b.i.d. = twice daily.) includes data from patients randomized to receive the sequence of treatment with oral tablets of placebo (randomization/Day 1 through Week 24) followed by metformin. Beginning at Week 24, patients were switched in a blinded manner to active treatment with metformin administered as 500 mg q.d. (q.d. = once daily) increased over 4 weeks by increments of 500 mg per week to a stable dose of 1000 mg b.i.d. Patients in this group continued to take metformin 1000 mg b.i.d for the remainder of the up to 30-week Phase B base study treatment period and during the extension study of up to 50 weeks.
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 175 | 178 | 177 | 183 | 178 | 165
Percent | -0.66 [-0.83 to -0.50] | -0.82 [-0.98 to -0.66] | -1.13 [-1.29 to -0.97] | -1.40 [-1.56 to -1.24] | -1.90 [-2.06 to -1.74] | 0.17 [0.00 to 0.33]

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 178 | 179 | 179 | 183 | 180 | 169
mg/dL | -17.5 [-24.1 to -10.8] | -27.3 [-34.0 to -20.7] | -29.3 [-35.9 to -22.6] | -47.1 [-53.7 to -40.6] | -63.9 [-70.5 to -57.3] | 5.8 [-1.0 to 12.7]

3. Secondary Outcome: Change From Baseline in 2-Hour PMG (Post-Meal Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 136 | 141 | 138 | 147 | 152 | 129
mg/dL | -51.9 [-62.3 to -41.5] | -53.4 [-63.6 to -43.2] | -78.0 [-88.3 to -67.6] | -92.5 [-102.6 to -82.5] | -116.6 [-126.4 to -106.7] | 0.3 [-10.4 to 11.0]

4. Secondary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 54
Description: HbA1c is measured as a percent. This change from baseline reflects the Week 54 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Week 54
Population: The Phase B Full Analysis Set (BFAS) included all patients with a baseline value and ≥1 value in Phase B (post-Week 24) for this outcome. Data following glycemic rescue were treated as missing. For BFAS patients with no data at Week 54, the last observed measurement was carried forward to Week 54.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 106 | 117 | 134 | 147 | 153 | 78
Percent | -0.82 [-1.00 to -0.63] | -1.01 [-1.18 to -0.83] | -1.34 [-1.50 to -1.17] | -1.41 [-1.57 to -1.25] | -1.80 [-1.96 to -1.65] | -1.10 [-1.32 to -0.88]

5. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 54
Description: Change from baseline at Week 54 is defined as Week 54 minus Week 0.
Time Frame: Week 54
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 105 | 117 | 134 | 146 | 153 | 78
mg/dL | -16.0 [-23.2 to -8.7] | -29.0 [-35.9 to -22.2] | -39.6 [-46.0 to -33.2] | -42.5 [-48.6 to -36.3] | -55.6 [-61.6 to -49.6] | -43.9 [-52.3 to -35.5]

6. Secondary Outcome: Change From Baseline in 2-Hour PMG (Post-Meal Glucose) at Week 54
Description: Change from baseline at Week 54 is defined as Week 54 minus Week 0.
Time Frame: Week 54
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 87 | 92 | 116 | 121 | 132 | 66
mg/dL | -45.9 [-57.2 to -34.6] | -58.6 [-69.6 to -47.6] | -76.3 [-86.1 to -66.5] | -89.6 [-99.2 to -80.0] | -107.9 [-117.1 to -98.7] | -80.9 [-93.9 to -67.9]

7. Secondary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 104
Description: HbA1c is measured as a percent. This change from baseline reflects the Week 104 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Week 104
Population: The Extension Full Analysis Set (EFAS) included all patients with a baseline value and ≥1 value in the extension (post-Week 54) for this outcome. Data following glycemic rescue were treated as missing. For EFAS patients with no data at Week 104, the last observed measurement was carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 50 | 64 | 87 | 96 | 105 | 42
Percent | -1.15 [-1.37 to -0.92] | -1.06 [-1.26 to -0.87] | -1.34 [-1.51 to -1.17] | -1.39 [-1.55 to -1.22] | -1.66 [-1.81 to -1.50] | -1.39 [-1.63 to -1.15]

8. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 104
Description: Change from baseline at Week 104 is defined as Week 104 minus Week 0.
Time Frame: Week 104
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 50 | 63 | 87 | 96 | 105 | 41
mg/dL | -26.8 [-36.2 to -17.4] | -41.4 [-49.8 to -33.0] | -43.2 [-50.3 to -36.2] | -47.5 [-54.3 to -40.7] | -57.3 [-63.7 to -50.8] | -45.2 [-55.7 to -34.8]

9. Secondary Outcome: Change From Baseline in 2-Hour PMG (Post-Meal Glucose) at Week 104
Description: Change from baseline at Week 104 is defined as Week 104 minus Week 0.
Time Frame: Week 104
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d.
Number analyzed (Participants) | 40 | 49 | 69 | 78 | 88 | 31
mg/dL | -74.1 [-90.3 to -57.9] | -72.7 [-87.4 to -58.1] | -86.7 [-99.0 to -74.5] | -96.2 [-107.8 to -84.6] | -110.0 [-120.9 to -99.1] | -93.3 [-111.8 to -74.9]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC
Serious Adverse Events (participants affected / at risk) | 15 | 10 | 14 | 17 | 13 | 23 | 3
Other Adverse Events (participants affected / at risk) | 71 | 74 | 99 | 87 | 94 | 73 | 40
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC
Any Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Cardiac Disorders (Cardiac disorders) | 2/179 | 1/182 | 3/182 | 3/190 | 3/182 | 4/176 | 0/117
Acute Coronary Syndrome (Cardiac disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 1/182 | 0/176 | 0/117
Acute Myocardial Infarction (Cardiac disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Angina Pectoris (Cardiac disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Angina Unstable (Cardiac disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Cardiac Failure (Cardiac disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Coronary Artery Disease (Cardiac disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 3/176 | 0/117
Myocardial Infarction (Cardiac disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 2/182 | 0/176 | 0/117
Myocardial Ischaemia (Cardiac disorders) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Palpitations (Cardiac disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Congenital, Familial And Genetic Disorders (Congenital, familial and genetic disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Exomphalos (Congenital, familial and genetic disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Any Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Vertigo Positional (Ear and labyrinth disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 1/179 | 0/182 | 1/182 | 1/190 | 2/182 | 2/176 | 0/117
Abdominal Hernia (Gastrointestinal disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Gastritis (Gastrointestinal disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Intestinal Obstruction (Gastrointestinal disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Pancreatitis Acute (Gastrointestinal disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 1/176 | 0/117
Swollen Tongue (Gastrointestinal disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any General Disorders And Administration Site Conditions (General disorders) | 0/179 | 1/182 | 0/182 | 3/190 | 0/182 | 3/176 | 0/117
Death (General disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Hernia Obstructive (General disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Non-Cardiac Chest Pain (General disorders) | 0/179 | 1/182 | 0/182 | 2/190 | 0/182 | 1/176 | 0/117
Sudden Cardiac Death (General disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any Hepatobiliary Disorders (Hepatobiliary disorders) | 0/179 | 1/182 | 1/182 | 0/190 | 0/182 | 3/176 | 0/117
Cholangitis Acute (Hepatobiliary disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Cholecystitis (Hepatobiliary disorders) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Cholelithiasis (Hepatobiliary disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 2/176 | 0/117
Any Immune System Disorders (Immune system disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Anaphylactic Reaction (Immune system disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any Infections And Infestations (Infections and infestations) | 3/179 | 2/182 | 1/182 | 1/190 | 3/182 | 4/176 | 1/117
Arthritis Infective (Infections and infestations) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Bronchitis (Infections and infestations) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Cellulitis (Infections and infestations) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Diabetic Foot Infection (Infections and infestations) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Diverticulitis (Infections and infestations) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Erysipelas (Infections and infestations) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Perineal Abscess (Infections and infestations) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Peritonsillar Abscess (Infections and infestations) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Pneumonia (Infections and infestations) | 1/179 | 0/182 | 0/182 | 1/190 | 2/182 | 0/176 | 1/117
Scrotal Abscess (Infections and infestations) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Sepsis (Infections and infestations) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 1/179 | 1/182 | 4/182 | 1/190 | 2/182 | 1/176 | 0/117
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Electric Shock (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Femur Fracture (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Hand Fracture (Injury, poisoning and procedural complications) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Meniscus Lesion (Injury, poisoning and procedural complications) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Multiple Injuries (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Tendon Injury (Injury, poisoning and procedural complications) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Tendon Rupture (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Investigations (Investigations) | 0/178 | 0/181 | 0/181 | 0/188 | 1/181 | 0/172 | 0/115
Blood triglycerides increased (Investigations) | 0/163 | 0/171 | 0/170 | 0/182 | 1/171 | 0/158 | 0/107
Any Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 1/176 | 0/117
Gestational Diabetes (Metabolism and nutrition disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Ketoacidosis (Metabolism and nutrition disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0/179 | 1/182 | 1/182 | 1/190 | 2/182 | 0/176 | 0/117
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Arthritis (Musculoskeletal and connective tissue disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Back Pain (Musculoskeletal and connective tissue disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Neoplasms Benign, Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/179 | 3/182 | 2/182 | 2/190 | 1/182 | 4/176 | 1/117
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 0/182 | 1/190 | 1/182 | 1/176 | 1/117
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 1/182 | 0/190 | 0/182 | 0/176 | 0/117
Glomus Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 1/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Retroperitoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any Nervous System Disorders (Nervous system disorders) | 2/179 | 0/182 | 0/182 | 2/190 | 0/182 | 4/176 | 0/117
Cerebrovascular Accident (Nervous system disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Cervicobrachial Syndrome (Nervous system disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Paraesthesia (Nervous system disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Syncope (Nervous system disorders) | 1/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Thalamic Infarction (Nervous system disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Transient Ischaemic Attack (Nervous system disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 1/176 | 0/117
Any Renal And Urinary Disorders (Renal and urinary disorders) | 1/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Hydronephrosis (Renal and urinary disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Micturition Urgency (Renal and urinary disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Any Reproductive System And Breast Disorders (Reproductive system and breast disorders) | 1/179 | 0/182 | 0/182 | 1/190 | 1/182 | 0/176 | 0/117
Adenomyosis (Reproductive system and breast disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 1/182 | 0/176 | 0/117
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
Menorrhagia (Reproductive system and breast disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Any Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/179 | 0/182 | 0/182 | 1/190 | 0/182 | 0/176 | 0/117
Any Vascular Disorders (Vascular disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 1/117
Peripheral Vascular Disorder (Vascular disorders) | 0/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 1/117
Varicose Vein (Vascular disorders) | 1/179 | 0/182 | 0/182 | 0/190 | 0/182 | 0/176 | 0/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg q.d. | Metformin 500 mg b.i.d. | Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d. + Metformin 500 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. | Placebo/Metformin 1000 mg b.i.d. | Sitagliptin 50 mg b.i.d + Metformin 1000 mg b.i.d. OLC
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 19/179 | 23/182 | 42/182 | 31/190 | 35/182 | 17/176 | 18/117
Constipation (Gastrointestinal disorders) | 9/179 | 6/182 | 6/182 | 7/190 | 3/182 | 3/176 | 5/117
Diarrhoea (Gastrointestinal disorders) | 8/179 | 14/182 | 23/182 | 19/190 | 25/182 | 12/176 | 10/117
Nausea (Gastrointestinal disorders) | 2/179 | 6/182 | 19/182 | 10/190 | 12/182 | 4/176 | 7/117
Any Infections And Infestations (Infections and infestations) | 40/179 | 44/182 | 53/182 | 54/190 | 60/182 | 37/176 | 19/117
Bronchitis (Infections and infestations) | 3/179 | 3/182 | 10/182 | 7/190 | 20/182 | 8/176 | 3/117
Gastroenteritis (Infections and infestations) | 9/179 | 1/182 | 3/182 | 3/190 | 7/182 | 3/176 | 1/117
Influenza (Infections and infestations) | 8/179 | 11/182 | 14/182 | 11/190 | 9/182 | 5/176 | 3/117
Nasopharyngitis (Infections and infestations) | 11/179 | 9/182 | 11/182 | 10/190 | 9/182 | 11/176 | 6/117
Upper Respiratory Tract Infection (Infections and infestations) | 12/179 | 17/182 | 20/182 | 21/190 | 24/182 | 13/176 | 4/117
Urinary Tract Infection (Infections and infestations) | 0/179 | 8/182 | 13/182 | 11/190 | 8/182 | 4/176 | 3/117
Fasting blood glucose increased (Investigations) | 8/178 | 3/180 | 1/181 | 0/186 | 1/181 | 11/171 | 0/115
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 16/179 | 20/182 | 21/182 | 19/190 | 25/182 | 13/176 | 6/117
Arthralgia (Musculoskeletal and connective tissue disorders) | 7/179 | 7/182 | 11/182 | 7/190 | 13/182 | 3/176 | 3/117
Back Pain (Musculoskeletal and connective tissue disorders) | 9/179 | 9/182 | 7/182 | 11/190 | 13/182 | 9/176 | 1/117
Any Nervous System Disorders (Nervous system disorders) | 9/179 | 13/182 | 20/182 | 17/190 | 19/182 | 10/176 | 4/117
Dizziness (Nervous system disorders) | 3/179 | 5/182 | 11/182 | 2/190 | 8/182 | 3/176 | 1/117
Headache (Nervous system disorders) | 6/179 | 9/182 | 12/182 | 15/190 | 12/182 | 7/176 | 3/117

LIMITATIONS AND CAVEATS:
Non-serious adverse experience results represent those events included in the primary safety analysis for this study (i.e., events that occurred prior to the initiation of glycemic rescue therapy).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.